CLINICAL TRIAL: NCT02160522
Title: Endotracheal Tube Cuff Pressure in the Pediatric Emergency Department: A Pilot Study
Brief Title: Endotracheal Tube (ETT) Cuff Pressure Study in the Emergency Department (ED)
Status: Completed | Type: Observational
Sponsor: Edward Ferenczy (Other)
Responsible Party: Sponsor-Investigator, Edward Ferenczy, Emergency Medicine Fellow, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00215
Record Dates: First submitted 2014-05-23; First posted 2014-06-10 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Endotracheal Tube Cuff Pressure Pediatric Emergency
Keywords: Intubation; cuff; cuffed; endotracheal; tube; pressure; pediatric; child; children; emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cuffed ETT: Patients that are intubated with a cuffed endotracheal tube.
  Interventions: Device: Cuffed ETT

INTERVENTIONS:
Device: Cuffed ETT — Measurement of the cuff pressure on an endotracheal tube and lower pressure to a safe range if it is elevated.

SUMMARY:
Our study will measure the pressure of the endotracheal tube cuff in intubated patients in the emergency department.

DETAILED DESCRIPTION:
Although manometers are available for the purpose of measuring ETT intra-cuff pressures, they are not currently in use at our institution's Emergency Department. This prospective cohort study will endeavor to determine the incidence of unacceptably high ETT cuff pressures in the ED, laying the foundation for follow up studies on patient outcomes and the potential need for more careful management of intra-cuff pressures in the ED.

ELIGIBILITY:
Inclusion Criteria:

* cuffed ETT in place on arrival in the ED
* cuffed ETT placed while in the ED

Exclusion Criteria:

* ETT cuff electively left deflated by practitioner
* Uncuffed ETT used

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that are intubated with a cuffed endotracheal tube in the emergency department of Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Cuff pressure | One time in the ED prior to discharge to the ICU
  One measurement of the ETT cuff pressure after intubation in the emergency department.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ferenczy, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States